CLINICAL TRIAL: NCT00757653
Title: Retrieval Study and Histological Examination Of A Hip Femoral Components With Hydroxyapatite Coatings
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: slow enrollment
Sponsor: Zimmer Biomet (Industry)
Collaborators: Biomet U.K. Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BMET UK 04
Record Dates: First submitted 2008-09-22; First posted 2008-09-23 (Estimated); Last update posted 2017-06-20 (Actual); Status verified 2017-06

CONDITIONS: Femoral Neck Fractures
MeSH Terms: conditions — Femoral Neck Fractures

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- 1 (Active Comparator): Stem with plasma sprayed porous Titanium 6Al4V alloy + Plasma sprayed HA
  Interventions: Device: Hip stem with plasma sprayed porous Ti 6Al4V alloy + plasma sprayed HA
- 2 (Experimental)
  Interventions: Device: Hip stem with plasma spayed porous Titanium 6Al4V alloy + Bonemaster HA
- 3 (Active Comparator)
  Interventions: Device: Hip stem with Interloc Titanium surface + Bonemaster H.A

INTERVENTIONS:
Device: Hip stem with plasma sprayed porous Ti 6Al4V alloy + plasma sprayed HA — Hip stem with plasma sprayed porous Titanium 6Al4V alloy + plasma sprayed HA
  Arms: 1
Device: Hip stem with plasma spayed porous Titanium 6Al4V alloy + Bonemaster HA — Hip stem with plasma spayed porous Titanium 6Al4V alloy + Bonemaster HA
  Arms: 2
Device: Hip stem with Interloc Titanium surface + Bonemaster H.A — Hip stem with Interloc Titanium surface + Bonemaster H.A
  Arms: 3

SUMMARY:
Retrieval study and histological examination of BiMetric Femoral Components with hydroxyapatite coatings.

DETAILED DESCRIPTION:
A single type of femoral component with 3 different HA coatings will be evaluated in this study. Patients with fractured neck of femur requiring hemi-arthroplasty will be recruited. Safety and performance of the device will be determined by adverse events (device related or non-related), survival and histological exam.

ELIGIBILITY:
Inclusion Criteria:

* Fractured neck of femur requiring hemi-arthroplasty. Selection of subjects for this evaluation should include the following considerations:-.
* A likelihood of obtaining relief of pain and improved function.
* Full skeletal maturity.
* Ability to follow instructions.
* Good general health for age.
* Willing to return for follow-up evaluations .
* No bias to sex.

Exclusion criteria:

• None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 57 (Actual)
Dates: Start 2003-10; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
Adverse Event | Anytime

SECONDARY OUTCOMES:
Histological Exam | Anytime

CONTACTS AND LOCATIONS:
Overall Officials: Helmut Zahn, FRCS, Principal Investigator — William Harvey Hospital
Locations (1):
- William Harvey Hospital, Ashford, Kent, United Kingdom